CLINICAL TRIAL: NCT07168499
Title: D-SCAPE - Diet and Stress Management Combined With Advanced Therapy for Crohn's and Ulcerative Colitis - A Pragmatic Clinical Trial
Brief Title: Diet and Stress Management Combined With Advanced Therapy for Crohn's and Ulcerative Colitis
Acronym: D-SCAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ashwin Ananthakrishnan, Principal Investigator and Clinical Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025P001274
Record Dates: First submitted 2025-08-28; First posted 2025-09-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: IBD (Inflammatory Bowel Disease)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A - Combined diet + stress management (Active Comparator): Subjects will receive a visit with an IBD dietician and a visit with an IBD GI psychologist (whether in person or virtual) within the first month of advanced therapy initiation and another visit with each of the IBD dietician and the IBD GI psychologist 4+/- 2 weeks after first intervention visit.
  Interventions: Behavioral: Diet Management; Behavioral: Stress Management
- Group B - Diet Alone (Active Comparator): Subjects will receive a visit with an IBD dietician (whether in person or virtual) within the first month of advanced therapy initiation and another visit with the IBD dietician 4+/-2 weeks after first intervention visit. They will be later offered a visit with an IBD GI psychologist after 3 months (after assessment of our primary outcomes).
  Interventions: Behavioral: Diet Management
- Group C - Stress management alone (Active Comparator): Subjects will receive a visit with an IBD GI psychologist (whether in person or virtual) within the first month of advanced therapy initiation and another visit with the IBD GI psychologist 4+/-2 weeks after first intervention visit. They will be later offered a visit with an IBD dietician after 3 months (after assessment of our primary outcomes).
  Interventions: Behavioral: Stress Management
- Group D - Usual Care Arm (No Intervention): Subjects will be offered a visit with an IBD GI psychologist and IBD dietician (whether in person or virtual) after 3 months (after assessment of our outcomes).

INTERVENTIONS:
Behavioral: Diet Management — Visit with IBD dietician for diet management specifically for IBD
  Arms: Group A - Combined diet + stress management; Group B - Diet Alone
Behavioral: Stress Management — Visit with IBD GI psychologist for stress management
  Arms: Group A - Combined diet + stress management; Group C - Stress management alone

SUMMARY:
Inflammatory Bowel Disease (IBD), which includes Crohn's Disease (CD) and Ulcerative Colitis (UC), is a chronic, immune-mediated disease characterized by recurrent episodes of relapse. The goal of this single site, pragmatic, randomized trial is to answer if combining lifestyle modifications (mindfulness/stress management + nutrition support) with advanced therapies for induction and maintenance of clinical remission in CD and UC as evaluated by disease activity scores in patients with active CD and UC.

Researchers will compare 4 study arms (Group 1, Group 2, Group 3, and Group 4) to see if combining lifestyle modifications with advanced therapies for induction and maintenance will show improvement in condition as evaluated by disease activity scores.

Groups:

1. Group A - Subjects will receive a visit with an IBD dietician and a visit with an IBD GI psychologist within the first month of advanced therapy initiation and another visit with both parties 4+/-2 weeks after the first intervention visit.
2. Group B - Subjects will receive a visit with an IBD dietician within the first month of advanced therapy initiation and another visit 4+/-2 weeks after the first intervention visit. They will later be offered a visit with an IBD GI psychologist after 3 months (after assessment of our primary outcomes).
3. Group C - Subjects will receive a visit with an IBD psychologist within the first month of advanced therapy initiation and another visit with the IBD GI psychologist 4+/-2 weeks after the first intervention visit. They will later be offered a visit with an IBD dietician after 2 months (after assessment of our primary outcomes).
4. Group D - Subjects will be offered a visit with an IBD GI psychologist and IBD dietician after 3 months (after assessment of our primary outcomes).

All subjects will be asked to complete a set of questionnaires and have the option to give blood and stool samples throughout the life of their participation in the study at certain visits.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to screening and to comply with the requirements of the study protocol.
2. At least 18 years of age
3. Established diagnosis of CD, UC, or IBD-unspecified
4. Recent (within 6 months) objective evidence of active IBD on colonoscopy or intestinal ultrasound or cross-sectional imaging or elevated inflammatory markers (CRP)
5. Initiating advanced therapy (anti-TNF agents, anti-integrin agents, anti-IL12/23, anti-IL23 agents, S1P receptor modulators, JAK inhibitors) for IBD per usual clinical care within 2 weeks of baseline/randomization, regardless of prior exposure to advanced therapies or disease duration
6. Other non-biologic IBD medications must remain stable during the treatment period and no medication changes are planned with the exception of tapering of corticosteroids.
7. Current disease activity defined as a Harvey Bradshaw index > 4 at baseline (week 0) for CD subjects or Simple Clinical Colitis Activity Index > 2 at baseline (week 0) for UC subjects or having had a recent exacerbation being treated with systemic steroids or budesonide.

Exclusion Criteria:

1. Inability to provide informed consent or unwilling or unlikely to comply with the requirements of the study.
2. Initiation of advanced therapy for extra-intestinal symptoms alone
3. Known eating disorders
4. Already receiving dietary therapy or stress management interventions
5. Severe untreated psychiatric comorbidity including history of suicidal thoughts
6. Evidence of untreated infection (e.g. Clostridium difficile)
7. Presence of stoma or J-pouch
8. Female subjects who are pregnant, lactating, or intending to become pregnant during the study period
9. On total parental nutrition (TPN) or already following a therapeutic diet for IBD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Change marked by clinical remission of IBD | 12 weeks, 24 weeks
  Subjects in the intervention arms will show clinically significant improvement in IBD symptoms after week 12 of the treatment period based upon disease activity scores using the Harvey-Bradshaw Disease Activity Index (HBI). For the HBI, a score less than 3 indicates remission while a score of 8-9 reflects severe disease.

SECONDARY OUTCOMES:
Clinical responses | 12 weeks, 24 weeks
  A secondary objective is to evaluate if clinical response to medications is changed with the interventions as measured by the HBI disease activity index.
Change in patient illness perception about disease and self-reported outcomes | 12 weeks, 24 weeks
  Subjects in the intervention arms will show clinically significant improvement in perception of IBD illness and self-reported outcomes after week 12 of the treatment period based upon Brief Illness Perception Questionnaire (B-IPQ) and Patient-Reported Outcomes Measurement Information System for Depression and Anxiety. For the B-IPQ, the lowest score is 0 and the highest is 10, with 10 indicating poorer overall view of illness. For both PROMIS questionnaires, a minimum score of 55 is within normal limits while scores above 70 are labelled as "severe."

OTHER OUTCOMES:
Evaluate the effect of intervention on change in fecal calprotectin levels between baseline and 12 weeks | 12 weeks
  Fecal calprotein will be measured using standardized testing to assess levels at baseline and at 12 weeks to see if there is a change in levels.
Change in levels of blood tests | 12 weeks
  Blood tests will be taken as part of standard of care and assessed for CBC with differential, comprehensive metabolic panel, C-reactive protein, ESR, serum iron studies, vitamin B12 level and processed for metagenomics to assess for changes post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Ananthakrishnan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided